CLINICAL TRIAL: NCT05883007
Title: Safety Cohort Study for Dose Optimization of Accelerator-based BPA-BNCT in Patients With Unresectable Locally Recurrent Squamous Cell Carcinoma of the Head and Neck (ST-BNCT2001)
Brief Title: Dose Optimized BNCT for Head and Neck Cancer
Acronym: ST-BNCT2001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Tohoku BNCT Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-BNCT2001
Record Dates: First submitted 2023-05-16; First posted 2023-05-31 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-optimized BNCT with borofalan(10B) (Experimental)
  Interventions: Radiation: Accelerator-based BNCT with borofalan(10B)

INTERVENTIONS:
Radiation: Accelerator-based BNCT with borofalan(10B) — Patients will be treated with BNCT regulated as 12, 15, or 18 Gy-Eq of the mucosal maximum dose.

SUMMARY:
The goal of this clinical trial is to evaluate the safety of applying BNCT with the dose optimization in patients with recurrent head and neck cancer. The main questions it aims to answer are:

- Dose optimized BNCT are conducted safety in these patients. Participants will receive dose optimized BNCT regulated as 12, 15, 18 Gy-Eq of the mucosal dose.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent to participate in the clinical trial on their own free will.
* Aged over 20 years at the time of consent obtaining.
* ECOG performance status (PS) of 0-2.
* Histologically confirmed a primary lesion of Head and Neck cancer.
* Following condition:

  1. Locally Recurrent Head and Neck Squamous Cell Carcinoma after chemo radiotherapy or radiation therapy.
  2. Primary Head or Neck Squamous Cell Carcinoma with no indicated of radical radiation therapy for the target lesions.
* More than one the target lesions based on RECIST (version 1.1)
* Local recurrent lesion localized to unilateral.
* Received a fractionated radiation therapy with total doses of ≥40 and ≤80 Gy at around 2 Gy per daily fraction at target lesion sites or an equivalent biologically effective dose.
* ≥50 days have passed since the last irradiation date of the prior radiation therapy at target lesion sites to the day of scheduled BNCT
* Have an estimated survival of ≥90 days after BNCT.
* Estimated able to receive the minimum tumor dose at least 20Gy-Eq.
* Screening test values that meet the following criteria.
* No abnormal findings of clinical concern in chest X-ray exam.

Exclusion Criteria:

* Active multiple primary cancers.
* Distant metastatic lesions.
* Active infections requiring systemic treatment.
* Serious complications.
* Poorly controlled diabetes mellitus.
* Poorly controlled hypertension.
* Chronic lung diseases.
* Kidney diseases.
* Cardiac diseases.
* Other serious complications.
* Phenylketonuria.
* Hereditary fructose intolerance.
* Current or past medical history of serious hypersensitivity to drugs or contrast media.
* Myocardial infarction, unstable angina, or poorly controlled arrhythmia within 6 months prior to the scheduled BNCT.
* Grade ≥3 (CTCAE v4.0) symptom at the target site.
* Tumor invasion of the carotid artery or adjacent to over half of the carotid artery.
* Dental caries whose treatment has not been completed.
* Received antitumor drugs within 4 weeks prior to the scheduled BNCT.
* Participating in a clinical study of an unapproved drug except 18F-F BPA-PET/CT examinations within 4 weeks prior to the scheduled BNCT.
* Implanted with a cardiac pacemaker, ventricular assist device, or the like.
* Inability to immobilize at a right position during irradiation by the investigator (subinvestigator)
* Pregnant or who are breastfeeding during the period of the clinical trial.
* Mental illness or mental conditions.
* Poorly controlled epilepsy.
* Unable to comply with the protocol and to attend follow-up visits.
* With a history of BNCT.
* Considered unfit to participate in this clinical trial as assessed by the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (Absence and presence of serious adverse events) | Within 90days after the completion of BNCT
  Grade 3 or higher adverse events as evaluated in CTCAEv5.1 Number of participants with severe adverse events due to an excess of tissue tolerance dose

SECONDARY OUTCOMES:
Objective response rate: ORR | Within 90 days after the completion of BNCT
  ORR within 90 days after the completion of BNCT is evaluated using RECIST guidelines (version 1.1).
  ORR is defined as the percentage of subjects with CR and PR in the target lesions among all eligible subjects.
Duration of Response | Within 2 years after the completion of BNCT
  The duration of the response is the time from the confirmed achievement of CR or PR (whichever is recorded first) to the date of initial objectively confirmed recurrence or exacerbation.
Disease control rate (DCR) | Within 90 days after the completion of BNCT
  DCR is evaluated using RECIST guidelines (version 1.1). DCR is defined as the proportion of subjects with CR, PR, or SD in the target lesions among all eligible subjects.
Overall survival (OS) | Within 2 years after the completion of BNCT or up to the end of this study
  OS is defined as the time from the day of the completion of BNCT to death due to all causes. The survey period will be up to the completion of the follow-up survey for all subjects.
Progression-Free Survival (PFS) | Within 2 years after the completion of BNCT or up to the end of this study
  PFS is defined as the time from the day of the completion of BNCT to the date of initial confirmed PD. The survey period will be up to the completion of the follow-up survey for all subjects.
Late Adverse Events | From 90 days to 2 years after the completion of BNCT
  The late Adverse Events are defined as the medical occurrence of the study from the treatment periods to the follow-up periods.
Quality of life (QOL) Score Based on EORTC QLQ C30 and H&N35. | Within 2 years after the completion of BNCT or up to the end of this study
  QOL score is assessed with EORTC QLQ C30 and H&N35 in the follow-up period. Results are scored as a specified manner by EORTC and changes in scores during the follow up period are evaluated
Quality-Adjusted Life Year (QALY) | Within 2 years after the completion of BNCT or up to the end of this study
  QOL and life year are multiplied to calculate the QALY. QOL score based on EQ-5D-5L in Japanese version.

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Tohoku BNCT Research Center, Kōriyama, Fukushima, Japan

IPD SHARING:
Plan to Share IPD: No